CLINICAL TRIAL: NCT05560620
Title: Impact of Sleep Deprivation on Objective, Physiological Measures of Brain Function Cognition
Brief Title: Sleep Deprivation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeuroCatch Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: NCI_NCClin_006
Record Dates: First submitted 2022-06-07; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Cognitive Change; Sleep Deprivation; Caffeine
MeSH Terms: conditions — Sleep Deprivation | interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: 2-group, randomized design
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sleep Deprivation and Caffeine Intervention (Experimental): Participants randomized into the sleep deprivation group and then randomized into receiving caffeinated coffee the next morning. Participant is blinded to the caffeine intervention.
  Interventions: Behavioral: Sleep Deprivation; Other: Caffeine
- Sleep Deprivation and no Caffeine intervention (Sham Comparator): Participants randomized into the sleep deprivation group and then randomized into receiving de-caffeinated coffee the next morning. Participant is blinded to the caffeine intervention.
  Interventions: Behavioral: Sleep Deprivation; Other: No Caffeine
- Control and Caffeine (Active Comparator): Participants randomized into the control group, who will sleep regularly, and then randomized into receiving caffeinated coffee the next morning. Participant is blinded to the caffeine intervention.
  Interventions: Other: Caffeine
- Control and No Caffeine (Sham Comparator): Participants randomized into the control group, who will sleep regularly, and then randomized into receiving de-caffeinated coffee the next morning. Participant is blinded to the caffeine intervention.
  Interventions: Other: No Caffeine

INTERVENTIONS:
Behavioral: Sleep Deprivation — Participants will be randomized into either the sleep deprivation group or the control group, who will sleep regularly.
  Arms: Sleep Deprivation and Caffeine Intervention; Sleep Deprivation and no Caffeine intervention
Other: Caffeine — On Day 2 morning, after the sleep deprivation or sleeping, participants will be randomized into receiving caffeinated or de-caffeinated coffee, which they will be blinded to.
  Arms: Control and Caffeine; Sleep Deprivation and Caffeine Intervention
Other: No Caffeine — De-caffeinated coffee
  Arms: Control and No Caffeine; Sleep Deprivation and no Caffeine intervention

SUMMARY:
The purpose of this study is to evaluate the measures of brain function, both neurophysiological (event-related potentials (ERPs) and functional (cognitive assessments), in response to sleep deprivation.

ELIGIBILITY:
Inclusion Criteria:

1. Any sex, between the ages of 19 and 45.
2. Able to understand the informed consent form, study procedures and willing to participate in study
3. Able to perform the testing required by the study.
4. Able to remain seated for 10 minutes
5. In good health with no history of clinically relevant neurological illness, acute disease or conditions or injury in the last 5 years.
6. A score of ≤ 5 on the Pittsburgh Sleep Quality Index (PSQI)
7. A score between 42 and 58 on the Morningness- Eveningness Questionnaire (MEQ)
8. Coffee consumption of < 5 cups per day.
9. Alcohol consumption of <15 units per week.
10. Self-described regular sleep pattern for the last 2 weeks.
11. Willing to consume caffeine in coffee form
12. Follow regular daily routine 24 hours prior to Baseline and between Baseline 1 and Baseline 2 study visits (i.e. sleep time, caffeine consumption etc.)

Exclusion Criteria:

1. Alcohol or CBD or THC consumption 24 hours prior to baseline and during the study
2. Currently and regularly taking sleep medications or supplements or medications that effect sleep
3. Any health condition (e.g. chronic fatigue) that would prevent the subject from completing the required testing.
4. Undergoing chemotherapy or any form of intensive long-term therapy.
5. Recent (3 months) injury or other acute condition that required treatment with pain killers or analgesics.
6. History of chronic pain or chronic headache disorders, including migraines.
7. History of TBI or condition that affects the brain or CNS.
8. Currently diagnosed with major psychiatric disorders (schizophrenia, bipolar, depression, generalized anxiety disorder)
9. Diagnosed with any memory disorders.
10. Currently diagnosed with any sleeping disorders (e.g. sleep apnea, hypersomnia, insomnia, parasomnia etc.)
11. Recent (in the last 6 months) history of alcohol or substance misuse.
12. Travel across time zones in the last 2 weeks.
13. Late night or evening shift work in the last 2 weeks.
14. Vaccination for COVID-19 within the last 72 hours prior to baseline.
15. Currently experiencing Covid-19 symptoms, including: fever or chills, cough, tiredness/fatigue, headache, sore throat, muscle or body aches, new loss of taste or smell, congestion or runny nose, nausea or vomiting, diarrhea, difficulty breathing or shortness of breath, or chest pain.)
16. If female and of child-bearing potential: pregnant, suspected or planning to become pregnant or breast-feeding
17. Contraindications for the NeuroCatch Platform:

17.1. Requires use of hearing aids or a cochlear implant 17.2. Diagnosed with tinnitus that is currently active 17.3. Temporary damage to hearing (e.g. punctured ear drum). 17.4. Implanted pacemaker or implanted electrical stimulators 17.5. Metal or plastic implants in the skull, excluding dental/facial implants. 17.6. Exposed to an investigational drug or device 30 days prior to start in this study, or concurrent or planned use of investigational drug or device while enrolled in this study* 17.7. Not proficient in the English language 17.8. Diagnosed epilepsy or history of seizures 17.9. If female and of child-bearing potential: pregnant, suspected or planning to become pregnant or breast-feeding 17.10. Unhealthy scalp (apparent open wounds and/or bruised or weakened skin) 17.11. Allergy to EEG gel

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Change in NeuroCatch® Platform 2 (NCP2), event-related potentials (ERPs) Amplitudes | 2 days
  N100, P300 and N400 amplitude values
Change in NeuroCatch® Platform 2 (NCP2), event-related potentials (ERPs) Latencies | 2 days
  N100, P300 and N400 latency values
Change in Cogstate cognitive assessment Accuracy scores from Baseline, Baseline 2 and Study Visit 3 (post-intervention) | 2 days
  accuracy (% of correct responses) scores
Change in Cogstate cognitive assessment Reaction time scores from Baseline, Baseline 2 and Study Visit 3 (post-intervention) | 2 days
  reaction time (ms) scores

SECONDARY OUTCOMES:
Change in NeuroCatch® Platform 2 (NCP2), event-related potentials (ERPs) pre and post caffeine intervention | 1 day
  N100, P300 and N400 amplitude and latency values
Change in Cogstate cognitive assessment measures (Detection Test, Identification Test, One Card Learning, and One Back Task) from Baseline, Baseline 2 and Study Visit 3 (post-intervention) | 1 day
  Cogstate accuracy (% of correct responses) and reaction time (ms) scores
Safety Measures | 2 days
  Frequency, severity and type of AEs, ADEs, and DDs
Demographics | 1 day
Medical History | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- HealthTech Connex Centre for Neurology Studies, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided